CLINICAL TRIAL: NCT06932640
Title: Continuous Assessment of Cerebral Autoregulation in Subarachnoid Hemorrhage (SAH) Patients Using Cerebral Oximetry Index and Hemoglobin Volume Reactivity Index
Brief Title: Continuous Assessment of Brain Blood Perfusion in Subarachnoid Hemorrhage Patients Using Near-Infrared Spectroscopy (NIRS)
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Weifeng Song, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300014488; Pending (Other Grant/Funding Number: Edwards Lifesciences Corp.)
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Aneurysmal subarachnoid hemorrhage (SAH) patients: The study will be conducted on patients aged 18 to 89 years admitted to the Neurological Intensive Care Unit (ICU) with a Aneurysmal subarachnoid hemorrhage (SAH). The study will use near-infrared spectroscopy (NIRS) monitors (which is outside standard of care) and transcranial doppler (TCD, only when available and is standard of care) that will be attached to these patients. The data from these devices will be used solely for analysis after the patients have been discharged.
  Interventions: Device: - Non-Invasive Near-infrared Spectroscopy (NIRS) device (HEM1 with Foresight Elite Sensor)

INTERVENTIONS:
Device: - Non-Invasive Near-infrared Spectroscopy (NIRS) device (HEM1 with Foresight Elite Sensor) — Near-Infrared Spectroscopy (NIRS) monitors, provided by Edwards Lifesciences, is a monitoring technique. It will be connected to consented patients, automatically capturing brain oxygen as waveform output, and stored in Sickbay system. The NIRS is a non-invasive monitoring method, in which adhesive pads will be applied to forehead. 4 hours continuous monitoring will be recorded on day 1 after SAH (or on presence to NICU), then every three days from day 3 to day 14 (within the DCI window), to 1 to 2 recordings from day 15 to day 21.

SUMMARY:
The goal of this observational study is to continuously assess cerebral autoregulation in patients with subarachnoid hemorrhage (SAH) using cerebral oximetry index (COx) and hemoglobin volume reactivity index (HVx). The main question it aims to answer is: Whether optimal perfusion pressure is dynamic and changes with time in patients with SAH, and that autoregulation is disrupted in patients during the course of SAH, contributing to delayed cerebral ischemia (DCI).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 89 years who are admitted to the Neurological Intensive Care Unit (Neuro ICU) between March 2025 and December 2026 for aneurysmal subarachnoid hemorrhage (SAH).

Exclusion Criteria:

* Patients under 18 years old
* Prisoners
* Pregnant women
* Patients enrolled in concurrent ongoing interventional trial
* Students of UAB
* Employees of UAB
* Patients who undergoes frontal decompression surgery resulting bone flap deficit where NIRS monitoring pads could not be applied.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurological Intensive Care Unit (NICU) patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Lower Limit of Autoregulation (LLA) | 21 days
  Successful calculations of moving Lower Limit of Autoregulation (LLA) for all three algorithms

SECONDARY OUTCOMES:
Change of delayed cerebral ischemia (DCI) to the average LLA | 21 days
  Correlation of clinical course of delayed cerebral ischemia (DCI) to average LLA
Change in time under LLA | 21 days
  Correlation in time under LLA
Change in dose under LLA | 21 days
  Correlation in dose under LLA

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Song, M.D., Ph.D, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided